CLINICAL TRIAL: NCT04070924
Title: Surgical Dressings After Endoscopic Carpal Tunnel Release: A Randomized Controlled Trial
Brief Title: Surgical Dressings After Endoscopic Carpal Tunnel Release
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI has chosen to prioritize other studies at this time.
Sponsor: Chris Grandizio (Other)
Responsible Party: Sponsor-Investigator, Chris Grandizio, Attending Physician, Geisinger Clinic
Organization: Geisinger Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-0474
Record Dates: First submitted 2019-08-24; First posted 2019-08-28 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional post-operative bulky soft tissue dressing (Active Comparator): 1. Intraoperative: MAC-Local Anesthesia; Local anesthetic mixture will be distributed in both the subcutaneous tissue and within the carpal canal
  2. Postoperative: Non-opioid medications only; Conventional post-operative bulky soft tissue dressing (Xeroform, 4x4s, Webril, Ace Wrap; Worn until first postoperative visit)
  Interventions: Other: Conventional bulky soft tissue dressing
- Bandaid post-operative dressing (Experimental): 1. Intraoperative: MAC-Local Anesthesia; Local anesthetic mixture will be distributed in both the subcutaneous tissue and within the carpal canal
  2. Postoperative: Non-opioid medications only; Bandaid over incision (Patient given an edema glove to wear starting post-operative day 1; Dressing change be changed post-operative day 2 and as needed after that)
  Interventions: Other: Bandaid

INTERVENTIONS:
Other: Bandaid — Bandaid dressing
  Arms: Bandaid post-operative dressing
Other: Conventional bulky soft tissue dressing — Conventional bulky soft tissue dressing
  Arms: Conventional post-operative bulky soft tissue dressing

SUMMARY:
Carpal tunnel syndrome (CTS) is the most common compressive neuropathy in the upper extremity. While carpal tunnel release (CTR), both open (OCTR) and endoscopic (ECTR), is safe and effective, there are questions regarding the use of postoperative dressings after surgery. It is not currently known if dressing choices influence post-operative pain, function or patient satisfaction after ECTR. A less cumbersome dressing (bandaid) may allow patients to perform daily tasks with more ease after surgery. The purpose of this investigation is to compare postoperative pain scores and patient satisfaction after ECTR for patients treated with conventional post-operative bulky soft tissue dressings versus those treated with a bandaid after surgery. The hypothesis is that patients using a bandaid after surgery will have an easier time with functional tasks after surgery and that pain scores will not significantly differ between the two groups. Furthermore, this study aims to determine if there are differences in patient satisfaction, functional outcomes, complications, and unscheduled healthcare contact between these two groups. This will be a randomized, controlled investigation.

DETAILED DESCRIPTION:
Carpal tunnel syndrome (CTS) is the most common compressive neuropathy in the upper extremity. While carpal tunnel release (CTR), both open (OCTR) and endoscopic (ECTR), is safe and effective, there are questions regarding the use of postoperative dressings after surgery. With recent attention to the opioid epidemic, there have been increasing efforts to reduce narcotic usage postoperatively while still controlling expected postoperative pain. Recent authors have found that many patients, particularly older patients, do not require any opioid analgesia after CTR with 47% of men and 36% of women consuming no narcotics after CTR (CHAPMAN). Furthermore, while splints have historically been used after surgery, their need has recently been questioned (LOGLI). It is not currently known if dressing choices influence post-operative pain, function or patient satisfaction after ECTR. A less cumbersome dressing (bandaid) may allow patients to perform daily tasks with more ease after surgery.

The purpose of this investigation is to compare postoperative pain scores and patient satisfaction after ECTR for patients treated with conventional post-operative bulky soft tissue dressings versus those treated with a bandaid after surgery. The hypothesis is that patients using a bandaid after surgery will have an easier time with functional tasks after surgery and that pain scores will not significantly differ between the two groups. Furthermore, this study aims to determine if there are differences in patient satisfaction, functional outcomes, complications, and unscheduled healthcare contact between these two groups. This will be a randomized, controlled investigation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 years of age or older
2. Patients undergoing primary, elective, unilateral ECTR under monitored anesthesia care with local anesthesia.

Exclusion Criteria:

1. Patients undergoing ECTR as part of a worker's compensation case
2. Patients currently incarcerated
3. Subject who cannot read and speak English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-03 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-03-20 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale Pain Score | 0-12 months
  best 0-10 worst; continuous scale to measure current pain level

SECONDARY OUTCOMES:
Boston Carpal Tunnel Questionnaire | 0-12 months
  ranges from 1 to 5, with a higher score indicating greater disability; -specific measure of self-reported symptom severity and functional status
PROMIS Pain Interference | 0-12 months
  best 0-100 worst; measures the effects of a patient's pain on their daily activities and lifestyle
PROMIS Self-Efficacy Manage Symptoms | 0-12 months
  best 0-100 worst; measures a patient's ability to cope with their symptoms related to the procedure
PROMIS Upper Extremity | 0-12 months
  worst 0-100 best; measures physical function of upper extremities
QuickDASH | 0-12 months
  best 0-100 worst; functional outcome score for disabilities of the arm, shoulder, and hand
number of participants with unscheduled healthcare contact | 0-12 months
  unscheduled healthcare contact includes patient calls/messages, emergency room visits, or scheduled clinic visits
morphine equivalents | 0-12 months
  morphine equivalents consumed for post-operative pain control
number of participants with complications | 0-12 months
  complications after surgery including infection and delayed healing
Satisfaction with overall outcome | 0-12 months
  11 point Likert scale; worst 0-10 best
Satisfaction postoperative pain control | 0-12 months
  11 point Likert scale; worst 0-10 best
Satisfaction with the dressing | 0-12 months
  11 point Likert scale; worst 0-10 best
Grip Strength Measurement | 0-12 months
  Using Jamar Hand Dynamometer, in kilograms ranging from worst 0-90 best

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Grandizio, MD, Principal Investigator — Geisinger Clinic